CLINICAL TRIAL: NCT07056803
Title: Sex Related Outcomes in Oral vs. Subcutaneous Semaglutide in Type 2 Diabetes Mellitus: A 12-month Real-world Study
Brief Title: Oral vs. Subcutaneous Semaglutide in Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Valentina Guarnotta, Principal investigator, University of Palermo
Other Study IDs: 04
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- oral semaglutide: oral semaglutide
  Interventions: Drug: Oral semaglutide
- subcutaneous semaglutide: subcutaneous semaglutide
  Interventions: Drug: subcutaneous semaglutide

INTERVENTIONS:
Drug: Oral semaglutide — Starting dose 3 mg for a month, followed by 7 mg for a month increased up to 14 mg a month
  Groups: oral semaglutide
Drug: subcutaneous semaglutide — subcutaneous semaglutide can be started at 0,25 mg a week for a month, to be increased at 0,5 mg a week, up to 1 mg a week
  Groups: subcutaneous semaglutide

SUMMARY:
This real-world, comparative cohort study aims to evaluate the 12-month effectiveness of oral versus subcutaneous semaglutide in patients with type 2 diabetes mellitus (T2D), with a specific focus on sex-based differences in metabolic response. A total of 212 patients were enrolled and evenly assigned to either oral or subcutaneous semaglutide. The primary outcome was the change in HbA1c, while secondary outcomes included variations in weight, lipid profile, liver function, and hepatic steatosis index. Subcutaneous semaglutide resulted in greater improvements in HbA1c, weight, and LDL cholesterol in men, while women exhibited a more favorable hepatic response. These findings support the need for sex-specific considerations in T2D therapy personalization.

DETAILED DESCRIPTION:
emaglutide is a GLP-1 receptor agonist approved for the treatment of type 2 diabetes mellitus (T2D), available in both once-weekly subcutaneous and once-daily oral formulations. While both have demonstrated efficacy in phase 3 trials (SUSTAIN and PIONEER programs), real-world comparative data-particularly regarding sex-based differences in response-remain limited. This prospective, observational, real-world cohort study aims to compare the 12-month metabolic efficacy and hepatic effects of oral versus subcutaneous semaglutide in patients with T2D, with a specific focus on sex-disaggregated outcomes.

A total of 212 adult outpatients with T2D diagnosed for at least one year were consecutively recruited from the Endocrinology and Metabolism Unit, University Hospital of Palermo. Patients were assigned to either oral or subcutaneous semaglutide (n = 106 per group), based on drug availability and patient preference, not clinical criteria. Both groups were matched for sex.

Inclusion criteria were: age ≥18 years, T2D diagnosis ≥1 year, no prior use of GLP-1 RAs, and baseline HbA1c >6.5% (48 mmol/mol).

Exclusion criteria included: pregnancy, participation in other interventional studies, and known hypersensitivity to semaglutide.

Patients received semaglutide titrated according to label:

Oral group: 3 mg/day for 4 weeks, then 7 mg/day; up-titration to 14 mg/day permitted in case of inadequate glycaemic response.

Subcutaneous group: 0.25 mg/week for 4 weeks, then 0.5 mg/week; up-titration to 1 mg/week allowed based on clinical judgement.

Primary endpoint: change in HbA1c at 12 months. Secondary endpoints: changes in body weight, waist circumference, lipid profile (LDL, HDL, triglycerides), liver enzymes (GOT, GPT), hepatic steatosis index (HSI), fibrosis-4 index (FIB-4), neutrophil-to-lymphocyte ratio (NLR), and platelet-to-lymphocyte ratio (PLR). The presence and degree of diabetic microvascular complications (retinopathy, nephropathy) were also assessed using established criteria.

Biochemical analyses were performed using standard enzymatic and immunoturbidimetric methods. LDL-C was calculated via the Friedewald formula. All parameters were recorded at baseline and at 12-month follow-up. Differences from baseline were calculated (Δ values), and statistical analysis included Shapiro-Wilk test for normality, t-tests for between-group comparisons, and sex-stratified analyses.

At 12 months, subcutaneous semaglutide led to greater reductions in HbA1c, weight, waist circumference, and triglycerides in the overall cohort. Among men, subcutaneous administration was associated with significantly lower Δ_weight, Δ_HbA1c, and Δ_LDL compared to oral. In women, subcutaneous semaglutide led to significantly lower Δ_HSI and Δ_GOT values, indicating a more favorable hepatic profile. No significant differences were found between sexes in the oral group.

These findings suggest a clinically meaningful interaction between semaglutide formulation and biological sex in real-world settings. The injectable formulation appears more effective in improving cardiometabolic parameters in male patients, while women may experience greater hepatic benefits. This supports the need for a sex-specific and formulation-aware approach to the management of T2D with GLP-1 RAs.

The study was approved by the Ethics Committee of the University Hospital "Paolo Giaccone" (Protocol number: 04/2024). All participants provided written informed consent. The trial was conducted in accordance with the Declaration of Helsinki and Good Clinical Practice guidelines.

ELIGIBILITY:
Exclusion criteria:

* pregnancy
* known allergy or hypersensitivity to semaglutide
* participation in another clinical trial during the treatment period

Inclusion criteria:

* age over 18 years
* diagnosis of T2D at least one year before the recruitment
* no treatment with prior GLP-1 RA
* baseline HbA1c >6.5% (48 mmol/mol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study investigated a population of adult outpatients with T2D diagnosed for at least 1 year, followed at the Endocrinology and Metabolism Division of the University Hospital of Palermo
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with HbA1c change | From enrollment to 12 months
  assess the change in HbA1c in patients treated with oral vs. subcutaneous semaglutide both in the entire cohort of patients and stratified by sex, over a 12-month period

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Paolo Giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Yes
We will share all the data by a journal publication
Supporting Information: CSR